CLINICAL TRIAL: NCT05658341
Title: Evaluating Effectiveness of an Integrative Intervention Based on Physical Activity, Nutrition and Supportive Care to Improve Quality of Life of Breast Cancer Survivors: Protocol for a Pragmatic Cluster Randomized Trial and Embedded Qualitative Study
Brief Title: Program of Physical Activity, Nutrition and Supportive to Improve the Quality of Life of Breast Cancer Survivors
Acronym: ADA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Siel Bleu (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ADA
Record Dates: First submitted 2022-12-02; First posted 2022-12-20 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Quality of Life; Breast Cancer
Keywords: Adapted physical activity; Breast cancer survivors
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This will be a pragmatic two-arm (ADA intervention versus control/usual care) cluster randomized controlled trial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADA intervention (Experimental): The ADA intervention arm
  Interventions: Behavioral: ADA
- Usual Care (Active Comparator): The usual care arm
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: ADA — The 12-weeks program will include one-hour in adapted physical activity (APA), and a discussion on relaxation techniques and the undertaking of deep breathing exercises (making them APA+ sessions). A series of "minute for nutrition" short information sheets will be distributed at the end of each session.
  Two workshops on "living better after breast cancer" will also be offered: one on general mobility and the other on daily nutrition.
  Moreover, women will be asked to set personal challenges as a method of motivational reinforcement, and will also be called for motivational check-ins at least 3 times. Follow-up calls will allow for further individualization, motivation, and the reception of participants' concerns or remarks.
  Further, participants in the intervention group will have access to a dedicated internet space containing several documents and videos on topics of concern to patients during the post-treatment phase.
  Arms: ADA intervention
Behavioral: Usual Care — Participants in the control group will be offered weekly APA sessions for 12 weeks, these sessions are based on current practices within the Siel Bleu organization. Sessions' content is adapted to people who have been treated for (all types) cancer and are based on current recommendations.
  These sessions are commonly organized by Siel Bleu in hospitals, community groups or local committees of the national league against cancer organization.
  Arms: Usual Care

SUMMARY:
Despite it being one of the leading causes of cancer death among women, survival following a breast cancer diagnosis has greatly increased in high-income countries. However; this gave rise to a growing population of women living long after breast cancer with a diminished quality of life (QoL) due to the long-term effects of cancer and cancer treatment.

Exercise can improve QoL, fatigue, and other mental and physical health outcomes in this population, and is strongly recommended among breast cancer survivors, much like a healthy diet. However adherence in real-life to these recommendations is seldom satisfactory. Also, evidence regarding the effect and cost-effectiveness of concurrent healthy lifestyle behaviors compared to exercise alone is limited. Hence the need to develop pragmatic (evaluating the effectiveness of interventions in real-life conditions) theoretical-based customized interventions, which aim to improve uptake and instill long-term adherence of health lifestyle among breast cancer survivors.

ADA (Activité physique adaptée Doublée d'un Accompagnement spécifique post-cancer) is an integrative intervention based on physical activity, nutrition and supportive care. The interventions aims to improve breast cancer survivors' physical and mental health and instill long-term healthy behaviors.

Our study will be a pragmatic two-arm (ADA intervention versus control/usual care) cluster randomized controlled trial which examines the effectiveness of the ADA intervention program.

The primary endpoint will be health-related quality of life, as measured at 12-month after the start of the trial.

Several secondary outcomes will also be assessed; which include Physical activity level, relationship to food and self-efficacy.

The study aims to recruit 160 participants in total, divided into 20 activity groups (clusters) of 8 participants.

Primary analyses will be carried out on an intention to treat (ITT) basis, at both cluster and participant level. All statistical analysis will adjust for the clustering of patients within centers as a random effect.

The aim of this trial is to provide scientific evidence on the 'real-world' effectiveness of an easily generalizable trial, with clinically-significant outcomes, touching a growing number of cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* adult women who are between 18 and 72 years of age
* had a diagnosis of localized breast cancer of any type, and who have completed their treatment (surgery, chemotherapy, radiotherapy) within the last 15 months, or still undergoing hormone therapy or nearing the end of their Herceptin treatment.
* French-speaking
* covered by the French Social Security system or benefiting from a similar health insurance system

Exclusion Criteria:

* A cancer diagnosis other than breast cancer, or a relapse/metastasis of breast cancer, or generalized cancer,
* A medical contraindication to exercise (a medical certificate of absence of contraindication to the practice of physical activity will be required, as for all physical activity in community settings).
* Significant visual or auditory problems or behavioral problems that make it difficult to participate in group physical activity sessions.
* a plan of moving away from the study site.
* participating in another clinical trial
* Male sex

Ages: 18 Years to 72 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life | 12 months after the beginning of the intervention
  The primary endpoint will be the health-related quality of life, as measured by the FACIT-F global score. This score is based on the 27-items Functional Assessment of Cancer Therapy-General (FACT-G) scale ,and the 13-items fatigue subscale included in the FACIT-F. Higher score indicate better Quality of life.

SECONDARY OUTCOMES:
Physical, social, emotional, and functional well-being | At 3 months, 6 months, and 12 months after the beginning of the intervention
  measured separately by the FACT-G four different subscales. Higher score indicate better Quality of life.
Fatigue | At 3 months, and 6 months after the beginning of the intervention
  measured by the FACIT-F global score. This score is based on the 13-items fatigue subscale included in the FACIT-F.
Physical activity level | At 3 months, 6 months, and 12 months after the beginning of the intervention
  Measured with the short version of the International Physical Activity Questionnaire (IPAQ-SF).A higher IPAQ-SF score indicates a better physical activity level..
Motivation for physical activity Questionnaire-2 (BREQ-2) scale | At 3 months, 6 months, and 12 months after the beginning of the intervention
  assessed with the short form of Behavioral Regulation in Exercise Questionnaire-2 (BREQ-2). A higher BREQ-2 score indicates a better exercise motivation.
Sedentary behavior (sitting time) | At 3 months, 6 months, and 12 months after the beginning of the intervention
  measured with a questionnaire adapted from the Recent Physical Activity Questionnaire (RPAQ). A higher RPAQ score indicates a lower sedentary behavior level.
Relationship to food | At 3 months, 6 months, and 12 months after the beginning of the intervention
  Measured using a scale adapted from the Positive Eating Scale. A Higher score indicates a positive relationship with eating.
Self-efficacy | At 3 months, 6 months, and 12 months after the beginning of the intervention
  people's beliefs about their ability to produce designated levels of performance that influence events that affect their lives, assessed by an ad-hoc scale

CONTACTS AND LOCATIONS:
Overall Officials: Gwenn Menvielle, PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France; Patricia Dargent, PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France; Fabienne El Khoury, PhD, Study Chair — Institut National de la Santé Et de la Recherche Médicale, France
Locations (8):
- France (8):
  - La Rochelle, La Rochelle, Charentes-maritimes
  - Saint Brieuc, Saint-Brieuc, Cotes d'Armor
  - Arpajon, Arpajon, Essonne
  - Brest, Brest, Finistere
  - Blagnac, Blagnac, Haute Garonne
  - Angers, Angers, Maine Et Loire
  - Pyrénées Atlantiques, Saint-Pée-sur-Nivelle, Pyrénées Atlantiques
  - La Roche sur Yon, La Roche-sur-Yon, Vendée

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El-Khoury F, Mino JC, Deschamps N, Lopez C, Menvielle G, Dargent-Molina P. Effectiveness of a community-based multicomponent lifestyle intervention (the ADA programme) to improve the quality of life of French breast cancer survivors: protocol for a pragmatic cluster randomised trial and embedded qualitative study. BMJ Open. 2024 Mar 14;14(3):e081447. doi: 10.1136/bmjopen-2023-081447. PMID 38485475